CLINICAL TRIAL: NCT00282776
Title: Identification and Therapy of Postpartum Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Wisner, Professor of Psychiatry, Obstetrics and Gynecology and Reproductive Sciences, Epidemiology and Women's Studies, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH071825 (NIH); R01MH071825 (NIH); DSIR 82-SEMS (Other: National Institute of Mental Health)
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Depression
Keywords: Postpartum Depression; Telephone Care Management; Screening for Postpartum Depression
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: TAU
- DCM (Experimental): Participants will receive care management for postpartum depression
  Interventions: Behavioral: Care Management for Postpartum Depression

INTERVENTIONS:
Behavioral: Care Management for Postpartum Depression — Depression Care Manager calls postpartum women and encourages women to seek appropriate depression care. In this context the depression care manager helps the women to identify barriers to appropriate care, her preferred method of care, and resources available. Calls are made initially at 2 calls per month, followed by one call per month and calls every other month for women who are doing well. Women assigned to this group receive research assessments at 3, 6, and 12 months postpartum. They also receive information about community and health plan resources available for women with depression.
  Arms: DCM
Behavioral: TAU — Participants receive treatment as usual for postpartum depression. Women assigned to this arm receive research assessments at 3, 6, and 12 months postpartum. At the baseline home visit where diagnostic assessments are completed women are given information about community and health plan resources if they choose to seek care for depression symptoms. Women are also given phone contact numbers for the research program.
  Arms: TAU

SUMMARY:
This study will evaluate the effectiveness of a telephone-based depression screening and care management program in treating depression in postpartum women.

DETAILED DESCRIPTION:
Depression is a serious illness that can interfere with everyday life. Researchers believe that it is one of the most common complications during and after pregnancy. Depression after pregnancy is called postpartum depression and may be caused by a rapid change in hormone levels during and immediately after pregnancy. Postpartum depression can occur anytime within the first year after childbirth and can negatively affect both mothers and their children. Mothers with postpartum depression may experience low energy, difficulty concentrating, irritability, and inability to meet their children's needs for love and affection. As a result, women with postpartum depression may feel guilty and lose confidence in themselves as parents. Research shows that children of mothers with postpartum depression may have delays in language development, difficulty with emotional bonding to others, behavioral problems, lower activity levels, sleep problems, and distress. This study will evaluate the effectiveness of a telephone-based depression screening and care management program in treating depression in postpartum women.

Participants in this single blind study will be randomly assigned to receive either enhanced treatment as usual or telephone-based care management for the first year postpartum. All participants will have a 90-minute in-home interview upon study entry to assess depressive symptoms, functional status, medical history, and post-pregnancy plans. Participants assigned to care management will receive two calls in the first month postpartum, followed by monthly calls for the remainder of the first postpartum year. During each 10- to 20-minute call, participants will be asked to provide information regarding current depressive symptoms, steps they have taken to seek depression-related care, and any barriers they have encountered in the process. In addition, a care manager will act as an advocate for the participants and assist in obtaining specialized services as necessary throughout the year. Participants assigned to receive enhanced treatment as usual will not receive monthly phone calls or tailored care management. All participants will receive follow-up calls at 3, 6, and 12 months postpartum to assess outcome measures; these calls will last about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 4-6 weeks postpartum
* English-speaking
* Score of at least 10 on the Edinburgh Postnatal Depression Scale

Exclusion Criteria:

* DSM-IV diagnosis of bipolar disorder or psychotic episode
* Active substance abuse within 6 months prior to study entry
* Has not received obstetrical care
* History of a suicide attempt within 6 months of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2006-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms, social functioning, and health | Measured at Months 3, 6, and 12 postpartum
Preferences for depression treatment | Measured at baseline and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Wisner, MD, RN, Principal Investigator — University of Pittsburgh
Locations (1):
- Women's Behavioral HealthCARE Program, Suite 410, 3501 Forbes Ave, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Burchfield TN, Yang A, Wisner KL, Clark CT. Rates of Major Depressive Disorder and Bipolar Disorder in Black and White Postpartum Women. J Clin Psychiatry. 2024 Nov 20;85(4):23m15023. doi: 10.4088/JCP.23m15023. PMID 39566056
- [Derived] Wisner KL, Sit DKY, McShea M, Luther JF, Eng HF, Dills JL, Moses-Kolko EL, Wisniewski SR. Telephone-Based Depression Care Management for Postpartum Women: A Randomized Controlled Trial. J Clin Psychiatry. 2017 Nov-Dec;78(9):1369-1375. doi: 10.4088/JCP.15m10563. PMID 28796940
- [Derived] Clark CT, Sit DK, Driscoll K, Eng HF, Confer AL, Luther JF, Wisniewski SR, Wisner KL. DOES SCREENING WITH THE MDQ AND EPDS IMPROVE IDENTIFICATION OF BIPOLAR DISORDER IN AN OBSTETRICAL SAMPLE? Depress Anxiety. 2015 Jul;32(7):518-26. doi: 10.1002/da.22373. Epub 2015 Jun 8. PMID 26059839
- [Derived] Wisner KL, Sit DK, McShea MC, Rizzo DM, Zoretich RA, Hughes CL, Eng HF, Luther JF, Wisniewski SR, Costantino ML, Confer AL, Moses-Kolko EL, Famy CS, Hanusa BH. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. JAMA Psychiatry. 2013 May;70(5):490-8. doi: 10.1001/jamapsychiatry.2013.87. PMID 23487258
- [Derived] Sit D, Seltman H, Wisner KL. Seasonal effects on depression risk and suicidal symptoms in postpartum women. Depress Anxiety. 2011 May;28(5):400-5. doi: 10.1002/da.20807. Epub 2011 Mar 4. PMID 21381158